CLINICAL TRIAL: NCT01703858
Title: An Open Label, Randomised, Single Dose, 3-way Cross Over Study to Investigate Relative Bioavailability and Food Effect on Different Formulations of BI 113608 in Healthy Male Subjects, Followed by Fixed Sequence Periods Investigating Influence of Pantoprazole Coadministration and Food Effect on Pharmacokinetics of Different Formulations of BI 113608
Brief Title: Study to Investigate the Relative Bioavailability, Influence of Pantoprazole Coadministration and Food Effect of Different Oral Formulation of BI 113608
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1314.3; 2012-002537-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (5):
- 1 BI 113608 (Active Comparator): powder in the bottle for oral solution, oral administration with 240 mL water
  Interventions: Drug: BI 113608 PIB
- 2 BI 113608 (Experimental): conventional tablet formulation
  Interventions: Drug: BI 113608
- 3 BI 113608 (Experimental): conventional tablet formulation, fed
  Interventions: Drug: BI 113608
- 4 BI 113608 (Experimental): conventional tablet after pantoprazole administration
  Interventions: Drug: pantoprazole 40 mg STADA; Drug: BI 113608
- 5 BI 113608 (Experimental): conventional tablet formulation, fasted, 0:30 min before fat breakfast
  Interventions: Drug: BI 113608

INTERVENTIONS:
Drug: BI 113608 PIB — powder for oral solution
  Arms: 1 BI 113608
Drug: BI 113608 — conventional tablet formulation
  Arms: 2 BI 113608
Drug: BI 113608 — conventional tablet formulation
  Arms: 3 BI 113608
Drug: BI 113608 — conventional tablet formulation
  Arms: 5 BI 113608
Drug: pantoprazole 40 mg STADA — film-coated tablet
  Arms: 4 BI 113608
Drug: BI 113608 — conventional tablet formulation
  Arms: 4 BI 113608

SUMMARY:
The objective of the trial is to investigate the relative bioavailability, influence of pantoprazole coadministration and food effect of different oral formulations of BI 113608 in healthy male subjects

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1314.3.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open label, randomised, single dose, 3-way cross-over study to investigate relative bioavailability and food effect on different formulations of Boehringer-Ingelheim (BI) -113608 in healthy male subjects, followed by fixed sequence periods investigating influence of pantoprazole coadministration and food effect on pharmacokinetics of BI-113608.
Groups:
- A - C - B - D - E: Participants first received single dose of oral solution of BI-113608 (50 milligram (mg)) under fasted conditions (A), then they received conventional tablet of BI-113608 (2 tablets of 25 mg) under fed conditions (C) and then the conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions (B) in 3-way crossover periods with washout phase of at least 6 days. After this participants received conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions following administration of pantoprazole 40 mg twice daily for 4 days with an additional 40 mg of pantoprazole 2 hours (h) prior to administration of BI-113608 (D) and then conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions 30 minutes (min) prior to a standardized high-calorie, high-fat breakfast (E). All doses were administered orally.
- B - A - C - D - E: Participants first received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions (B), then they received oral solution of BI-113608 (50 mg) under fasted conditions (A) and then the conventional tablet of BI-113608 (2 tablets of 25 mg) under fed conditions (C) in 3-way crossover periods with washout phase of at least 6 days. After this participants received conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions following administration of pantoprazole 40 mg twice daily for 4 days with an additional 40 mg of pantoprazole 2 h prior to administration of BI-113608 (D) and then conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions 30 min prior to a standardized high-calorie, high-fat breakfast (E). All doses were administered orally.
- C - B - A - D - E: Participants first received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fed conditions (C), then they received conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions (B) and then the oral solution of BI-113608 (50 mg) under fasted conditions (A) in 3-way crossover periods with washout phase of at least 6 days. After this participants received conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions following administration of pantoprazole 40 mg twice daily for 4 days with an additional 40 mg of pantoprazole 2 h prior to administration of BI-113608 (D) and then conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions 30 min prior to a standardized high-calorie, high-fat breakfast (E). All doses were administered orally.
Period: Overall Study
Arm/Group | A - C - B - D - E | B - A - C - D - E | C - B - A - D - E
Started | 5 | 5 | 5
Completed | 5 | 4 | 5
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All subjects those who received at least 1 dose of study drug were included in the in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | A - C - B - D - E | B - A - C - D - E | C - B - A - D - E | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (8.9) | 40.8 (8.6) | 41.8 (7.9) | 40.7 (7.9)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte BI-113608 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte BI-113608 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: PK plasma samples were taken at: 2 hours (h) before drug administration and 15 min, 30 min, 45 min, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 8h, 10h, 12h, 14h, 24h, 48h, 72h after drug administration.
Population: Pharmacokinetic (PK) set: It included all treated subjects who provided at least 1 observation for at least 1 primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol)* hours (h) / Litre (L)
Groups:
- A : BI-113608: Participants received single dose of oral solution of BI-113608 (50 milligram (mg)) under fasted conditions.
- B : BI-113608: Participants received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions orally.
- C : BI-113608: Participants received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fed conditions orally.
- D : BI-113608: Participants received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions orally following administration of pantoprazole 40 mg twice daily for 4 days with an additional 40 mg of pantoprazole 2 hours (h) prior to administration of BI-113608.
- E : BI-113608: Participants received single dose of conventional tablet of BI-113608 (2 tablets of 25 mg) under fasted conditions orally 30 minutes (min) prior to a standardized high-calorie, high-fat breakfast.
Arm/Group | A : BI-113608 | B : BI-113608 | C : BI-113608 | D : BI-113608 | E : BI-113608
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 14
nanomol (nmol)* hours (h) / Litre (L) | 936 (27.4) | 924 (31.2) | 648 (39.3) | 900 (32.7) | 759 (27.1)
Statistical Analysis 1: Comparison: A : BI-113608 vs B : BI-113608; B : BI-113608 vs. A : BI-113608 - Comparison with oral solution; Test type: Non-Inferiority or Equivalence — Assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratio of the geometric means (gMeans) with acceptance range of 80.00 to 125.00%; p = 0.0000, ANOVA; Relative bioavailability was estimated by the ratios of the adjusted geometric means. CIs were calculated based on the residual error; Ratio of Geometric means (%) = 98.68, 90% CI 2-sided [92.501 to 105.272], Standard Deviation 10.0 — Analysis of variance includes the effects: sequence, subjects nested within sequences, period and treatment in crossover; subject and treatment in fixed sequence. Standard deviation is actually Intra individual geometric coefficient of variation
Statistical Analysis 2: Comparison: B : BI-113608 vs C : BI-113608; C : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9644, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 70.16, 90% CI 2-sided [62.331 to 78.962], Standard Deviation 18.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: B : BI-113608 vs E : BI-113608; E : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2835, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 83.36, 90% CI 2-sided [73.648 to 94.346], Standard Deviation 18.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: C : BI-113608 vs E : BI-113608; E : BI-113608 vs. C : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1599, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 117.18, 90% CI 2-sided [104.923 to 130.867], Standard Deviation 16.7 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: B : BI-113608 vs D : BI-113608; D : BI-113608 vs. B : BI-113608 - Pantoprazole effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0020, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 97.40, 90% CI 2-sided [88.072 to 107.719], Standard Deviation 15.8 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Measured Concentration of the Analyte BI-113608 in Plasma (Cmax)
Description: Maximum measured concentration of the analyte BI-113608 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | A : BI-113608 | B : BI-113608 | C : BI-113608 | D : BI-113608 | E : BI-113608
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 14
nmol/L | 271 (44.6) | 242 (47.5) | 132 (77.8) | 196 (50.0) | 227 (53.1)
Statistical Analysis 1: Comparison: A : BI-113608 vs B : BI-113608; B : BI-113608 vs. A : BI-113608 - Comparison with oral solution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1261, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 89.26, 90% CI 2-sided [75.893 to 104.973], Standard Deviation 25.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: B : BI-113608 vs C : BI-113608; C : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9808, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 54.57, 90% CI 2-sided [40.711 to 73.157], Standard Deviation 47.4 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: B : BI-113608 vs E : BI-113608; E : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1449, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 94.88, 90% CI 2-sided [72.175 to 124.731], Standard Deviation 43.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: C : BI-113608 vs E : BI-113608; E : BI-113608 vs. C : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9463, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 169.46, 90% CI 2-sided [124.093 to 231.419], Standard Deviation 49.7 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: B : BI-113608 vs D : BI-113608; D : BI-113608 vs. B : BI-113608 - Pantoprazole effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4564, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 81.06, 90% CI 2-sided [65.811 to 99.848], Standard Deviation 33.3 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI-113608 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the analyte BI-113608 in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | A : BI-113608 | B : BI-113608 | C : BI-113608 | D : BI-113608 | E : BI-113608
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 14
nmol*h/L | 938 (27.4) | 926 (31.2) | 650 (39.3) | 902 (32.7) | 761 (27.1)
Statistical Analysis 1: Comparison: A : BI-113608 vs B : BI-113608; B : BI-113608 vs. A : BI-113608 - Comparison with oral solution; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 98.66, 90% CI 2-sided [92.500 to 105.225], Standard Deviation 9.9 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: B : BI-113608 vs C : BI-113608; C : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9635, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 70.24, 90% CI 2-sided [62.430 to 79.038], Standard Deviation 18.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: B : BI-113608 vs E : BI-113608; E : BI-113608 vs. B : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2771, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 83.46, 90% CI 2-sided [73.774 to 94.412], Standard Deviation 18.7 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: C : BI-113608 vs E : BI-113608; E : BI-113608 vs. C : BI-113608 - Food effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1584, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 117.16, 90% CI 2-sided [104.958 to 130.787], Standard Deviation 16.6 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: B : BI-113608 vs D : BI-113608; D : BI-113608 vs. B : BI-113608 - Pantoprazole effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0020, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric means (%) = 97.41, 90% CI 2-sided [88.066 to 107.741], Standard Deviation 15.8 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 14 days after the last drug administration, up to 42 days.
Groups:
- Pantoprazole 40mg: Participants received single dose of Pantoprazole 40mg alone twice daily for 4 days with an additional 40 mg of pantoprazole 2 hours (h) prior to administration of BI-113608.
Arm/Group | A : BI-113608 | B : BI-113608 | C : BI-113608 | Pantoprazole 40mg | D : BI-113608 | E : BI-113608
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 6/15 | 6/15 | 7/15 | 3/15 | 4/15 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A : BI-113608 (N=15) | B : BI-113608 (N=15) | C : BI-113608 (N=15) | Pantoprazole 40mg (N=15) | D : BI-113608 (N=15) | E : BI-113608 (N=14)
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 5 | 5 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes